CLINICAL TRIAL: NCT06457451
Title: Impact d'un Programme coordonné diététique-activité Physique adaptée Sur le Pourcentage de Masse Maigre d'Adultes Atteints de Mucoviscidose traités Par Elexacaftor-Tezacaftor-Ivacaftor : Essai contrôlé randomisé Multicentrique
Brief Title: Impact of a Coordinated Dietetic-adapted Physical Activity Program on the Percentage of Lean Body Mass in Adults With Cystic Fibrosis Treated With Elexacaftor-Tezacaftor-Ivacaftor: Multicentre Randomised Controlled Trial
Acronym: DIAPASOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: Fondation Ildys (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-A02715-40; DR220270 (Other: Sponsor)
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Cystic Fibrosis
Keywords: Elexacaftor-Tezacaftor-Ivacaftor; Cystic Fibrosis; Adapted Physical Activity; Body composition; Dietetic
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DIAPASOM program (Experimental): Program of adapted physical activity carried out remotely by a specialized instructor for one year:
  * Phase 1 (3 months): 2 supervised weekly sessions.
  * Phase 2 (3months): 1 supervised weekly session and 1 independent weekly session.
  * Phase 3 (6months): 2 independent weekly sessions with monthly telephone follow-up.
  Combined with personalized dietetic care by a dietician for one year too:
  In person dietetic consultation every 3 months to monitor personalized objectives, with telephone follow-up between each face-to-face consultation to improve compliance.
  Interventions: Other: DIAPASOM program
- Management as usual (No Intervention): Management of nutrition and physical activity as usual

INTERVENTIONS:
Other: DIAPASOM program — A program of adapted physical activity carried out remotely by a specialist instructor, combined with personalized dietetic care by a dietician for one year.
  Arms: DIAPASOM program

SUMMARY:
Cystic fibrosis is an autosomal recessive inherited disease linked to various mutations in the gene coding for the Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) protein, with respiratory and digestive disorders conditioning the prognosis.

Digestive damage may be responsible for malnutrition of multifactorial origin (insufficient energy intake, increased energy losses, increased basal metabolic rate), and studies show a correlation between reduced lean body mass and respiratory function.

In 2019, the French National Authority for Health (HAS) redefined undernutrition by including "quantified reduction in muscle mass and/or function" as a phenotypic diagnostic criterion.

Elexacaftor-Tezacaftor-Ivacaftor, an innovative therapy (authorization in 2021) for this population, aims to restore the function of CFTR protein. Significant improvements in lung function and weight gain were observed from the first weeks of treatment. These improvements have also led to the emergence of lesser-known nutritional problems in these patients, such as overweight and the development of metabolic complications. Nonetheless, new management options in terms of dietary adjustments and adapted physical activity for these patients are possible, given the development of their abilities.

Adapted Physical Activity (APA) helps to improve general muscular function by strengthening respiratory and skeletal muscles, improving aerobic capacity, and aiding bronchial drainage through muscle strengthening and endurance work. Maintaining or even increasing muscle mass depends not only on appropriate food intake and optimal dietary management, but also on regular physical activity, as recommended by the HAS.

Our hypothesis is therefore that a structured dietetic/adapted physical activity program (DIAPASOM program) can increase the percentage of lean body mass at 12 months in adult cystic fibrosis patients treated with Elexacaftor-Tezacaftor-Ivacaftor.

DETAILED DESCRIPTION:
Cystic fibrosis is an autosomal recessive inherited disease linked to various mutations in the gene coding for the Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) protein, with respiratory and digestive disorders conditioning the prognosis.

Digestive damage may be responsible for malnutrition of multifactorial origin (insufficient energy intake, increased energy losses, increased basal metabolic rate), and studies show a correlation between reduced lean body mass and respiratory function.

In 2019, the French National Authority for Health (HAS) redefined undernutrition by including "quantified reduction in muscle mass and/or function" as a phenotypic diagnostic criterion.

Elexacaftor-Tezacaftor-Ivacaftor, an innovative therapy (authorization in 2021) for this population, aims to restore the function of CFTR protein. Significant improvements in lung function and weight gain were observed from the first weeks of treatment. These improvements have also led to the emergence of lesser-known nutritional problems in these patients, such as overweight and the development of metabolic complications. Nonetheless, new management options in terms of dietary adjustments and adapted physical activity for these patients are possible, given the development of their abilities.

Adapted Physical Activity (APA) helps to improve general muscular function by strengthening respiratory and skeletal muscles, improving aerobic capacity, and aiding bronchial drainage through muscle strengthening and endurance work. Maintaining or even increasing muscle mass depends not only on appropriate food intake and optimal dietary management, but also on regular physical activity, as recommended by the HAS.

Our hypothesis is therefore that a structured dietetic/adapted physical activity program (DIAPASOM program) can increase the percentage of lean body mass at 12 months in adult cystic fibrosis patients treated with Elexacaftor-Tezacaftor-Ivacaftor.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 18 or over
* Suffering from cystic fibrosis
* Treated with Elexacaftor-Tezacaftor-Ivacaftor for at least 6 months
* Affiliated to a social security scheme
* with a signed Informed Consent form.

Exclusion Criteria:

* Pregnant and breast-feeding women
* Subject under legal protection, guardianship or curatorship
* Subject whose physical activity is not medically authorised or whose physical and motor capacities do not allow them to take part in physical activity.
* Subject who is unable to comply with the requirements of the DIAPASOM program
* Difficulty in understanding the self-questionnaires
* Wearing a pacemaker or metal prosthesis
* Fluid retention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Evolution of percentage of patients lean mass as a percentage of body mass | From randomization, up to 12 months
  Impedancemetry

SECONDARY OUTCOMES:
Evolution of percentage of patients fat mass as a percentage of body mass | From randomization, up to 12 months
  impedancemetry
Weight evolution | From randomization, up to 12 months
  Weight measurement
Body Mass Index (BMI) evolution | From randomization, up to 12 months
  Weight and height measurement
Cardio-respiratory endurance | From randomization, up to 12 months
  6-Minute Walk Test (6MWT)
Bilateral Handgrip strength | From randomization, up to 12 months
  Handgrip Test
Lower limb muscle power | From randomization, up to 12 months
  30-second Sit-to-Stand test
Upper limb muscle power | From randomization, up to 12 months
  Pump test
Static trunck extensors muscle endurance | From randomization, up to 12 months
  "Superman" test
Static trunck flexors muscle endurance | From randomization, up to 12 months
  Shirado-Ito test
Balance between static muscular endurance of extensors and flexors | From randomization, up to 12 months
  Calculated using the Shirado-Ito/"Superman" ratio
Posterior chain flexibility (Hamstring, hips and lower back) | From randomization, up to 12 months
  Front trunk flexion test
Upper limb flexibility | From randomization, up to 12 months
  scapulohumeral mobility test
Forced Expiratory Volume in 1 second (FEV1) | From randomization, up to 12 months
  Spirometry
Physical activity volume and sedentary time | From randomization, up to 12 months
  Physical activity and sedentary behavior self-questionnaire (ONAPS-PAQ)
Evolution of quality of life | From randomization, up to 12 months
  Cystic Fibrosis Questionnaire-Revised (CFQR-14)
Program feedback questionnaire | 12 months after randomization
  Self-questionnaire about how patients in the experimental group feel about the program

CONTACTS AND LOCATIONS:
Overall Officials: Julie MANKIKIAN, MD, Principal Investigator — University Hospital, Tours
Locations (4):
- France (4):
  - Cystic Fibrosis Resource and Competence Centre, University Hospital, Angers, Angers
  - Cystic Fibrosis Resource and Competence Centre, Fondation Ildys, Roscoff, Roscoff
  - Cystic Fibrosis Resource and Competence Centre, University Hospital, Tours, Tours
  - Cystic Fibrosis Resource and Competence Centre, Hospital, Tours, Vannes